CLINICAL TRIAL: NCT03093766
Title: Balance Study on ICU-acquired Hypernatremia and Sodium Handling
Brief Title: Balance Study on ICU-acquired Hypernatremia and Sodium Handling (BIAS)
Acronym: BIAS
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: ZRTPO 996
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2017-05

CONDITIONS: ICU-acquired Hypernatremia
Keywords: Aetiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to find differences between patients who do and do not develop ICU-acquired hypernatremia (IAH). Therefore extended sodium and fluid balances will be performed. Also a couple of other factors that possibly contribute to the development of IAH and/or could give clues about the mechanisms in the development of IAH will be investigated.

DETAILED DESCRIPTION:
ICU-acquired hypernatremia (IAH) is common in critically ill patients, but it's aetiology is still not fully understood. Sodium overload and inadequate fluid administration are generally considered important factors, but a previous retrospective study did not reveal differences in sodium or fluid balances between patients who did and did not develop IAH. Because this was retrospective these balances will be prospectively studied in this study to be more sure about the importances of these balances in the development of IAH. Previous studies indicated that (a lot) more factors contribute to the development of IAH. In this study these factors will be investigated, hoping to find differences between patients who do and do not develop IAH.

ELIGIBILITY:
Inclusion Criteria:

* Predicted duration of ICU-admission >48 hours

Exclusion Criteria:

* Renal replacement therapy
* Reason for admission necessitates actively elevation of serum sodium concentration
* Electrolyte disturbance as reason for admission
* ICU re-admission within 30 days
* Referral from another ICU
* Serum sodium concentration on admission 143mmol/l or above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All unplanned ICU-admissions
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Sodium balance | During ICU-admission
  Differences in sodium balances between patients who do and do not develop IAH
Fluid balance | During ICU-admission
  Differences in fluid balances between patients who do and do not develop IAH

SECONDARY OUTCOMES:
Kidney function | During ICU-admission
  Differences in parameters concerning kidney function (creatinine, urea) between patients who do and do not develop IAH
Inflammation | During ICU-admission
  Differences in inflammation (CRP, infections) between patients who do and do not develop IAH
Nutritional state | During ICU-admission
  Differences in nutritional state (albumin, BIVA-measurement) between patients who do and do not develop IAH

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Boerma, Principal Investigator — medical center leeuwarden
Locations (1):
- Medisch Centrum Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Collected data will be available through an online portal / storage website as soon as the manuscript was published. From that moment data can be obtained after a request via the online portal / storage website.

REFERENCES:
- [Background] Darmon M, Diconne E, Souweine B, Ruckly S, Adrie C, Azoulay E, Clec'h C, Garrouste-Orgeas M, Schwebel C, Goldgran-Toledano D, Khallel H, Dumenil AS, Jamali S, Cheval C, Allaouchiche B, Zeni F, Timsit JF. Prognostic consequences of borderline dysnatremia: pay attention to minimal serum sodium change. Crit Care. 2013 Jan 21;17(1):R12. doi: 10.1186/cc11937. PMID 23336363
- [Background] van IJzendoorn MC, Buter H, Kingma WP, Navis GJ, Boerma EC. The Development of Intensive Care Unit Acquired Hypernatremia Is Not Explained by Sodium Overload or Water Deficit: A Retrospective Cohort Study on Water Balance and Sodium Handling. Crit Care Res Pract. 2016;2016:9571583. doi: 10.1155/2016/9571583. Epub 2016 Sep 14. PMID 27703807
- [Background] Bihari S, Ou J, Holt AW, Bersten AD. Inadvertent sodium loading in critically ill patients. Crit Care Resusc. 2012 Mar;14(1):33-7. PMID 22404059